





## **Consent Form**

(Version: V 1.0, 28<sup>th</sup> March 2019)

Physiotherapy management Of urinary Incon Inence In athletic women (POsITIve) – a feasibility study

Phase 2: Physiotherapy for Urinary Incontinence

| Name of Researcher: | | |
|---|---|---|
| Dr ( | Gillian Campbell (Research Fellow, Daphne Jackson Trust), University of No | tingham |
| Naı | Name of Participant: | |
| 1. | I confirm that I have read and understand the information sheet version number V 1.0, dated 28/03/2019, for the above study and have had the opportunity to ask questions. | Please initial box |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, and without my legal rights being affected. I understand that should I withdraw then the information collected so far cannot be erased and that this information may still be used in the project analysis. | |
| 3. | I understand that the data collected in the study may be looked at by authorised individuals from the University of Nottingham, the research group, and regulatory authorities where it is relevant to my taking part in this study. I give permission for these individuals to have access to these records and to collect, store, analyse and publish information obtained from my participation in this study. I understand that my personal details will be kept confidential. | |

(Continued on following page)







| | | | Plea | ase initial box |
|---|---|---|---|---|
| 4. | I understand further, as part of my assessment and ongoing treatment, I will be asked to consent to a digital vaginal assessment of my pelvic floor muscles and their function. | | | |
| 5. | I understand that my data will be recorded throughout the intervention and may be used in the study reports. | | | |
| 6. | I understand that the information collected about me may be used to support other research in the future, and may be shared anonymously with other researchers. | | | |
| 7. | I agree to a courtesy letter regarding my participation in this study being sent to my GP | | | |
| 8. | I would like to know the results of the study and would like a summary of the findings to be sent to me once the study is complete.* | | | |
| 9. I agree to take part in the above study. | | | | |
| Nam | e of participant | Date | Signature | _ |
| Nam | e of person taking consent | Date | Signature | _ |

\* Contact details to be collected on separate sheet.

2 copies: 1 for participant, 1 for the project notes.